CLINICAL TRIAL: NCT02555423
Title: The Effects of Serratus Plane Block Performed Under Direct Vision on Post-operative Pain in Breast Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Kingston Hospital NHS Trust (Other)
Responsible Party: Principal Investigator, Marcus Hards, Doctor, Kingston Hospital NHS Trust
Purpose: Supportive Care
Other Study IDs: 179669
Record Dates: First submitted 2015-09-17; First posted 2015-09-21 (Estimated); Last update posted 2015-09-21 (Estimated); Status verified 2015-09

CONDITIONS: Post-operative Pain; Serratus Block; Breast Surgery
MeSH Terms: conditions — Pain, Postoperative

INTERVENTIONS:
Drug: Local anaesthetic - chirocaine

SUMMARY:
The aim of the study is to determine the effectiveness of serratus place block in the control of post-operative pain following mastectomy. The investigators will compare one group of patients receiving serratus plane block and wound infiltration to a control group receiving a saline injection into serratus anterior and wound infiltration with local anaesthetic only. The investigators will compare our results to the National Mastectomy and Breast Reconstruction Audit's reported rate of 6.2% of patients reporting severe pain following mastectomy to see if there is an improvement of the national standard. In the serratus block group, the investigators expect a 50% decrease in the number of patients who report severe pain day one post operatively.

DETAILED DESCRIPTION:
Patients who undergo mastectomy +/- sentinel node biopsy +/- axillary clearance +/- implant reconstruction will be eligible for the study. Patients will be consented by Mr Davies preoperatively in the breast clinic at Kingston Hospital to be randomly allocated to one of two groups.

The study will be double blinded and patients will be randomly allocated in to one of two groups as detailed below:

Group 1 - Control Group The first group will act as the control group and will receive wound infiltration with the full amount of local anaesthetic (40mls) around the drain sites and axillary wound, if present, as is standard practice. They will also receive a 20ml injection of 0.9% saline deep to serratus anterior under direct observation. Infiltration of saline will be delivered into 2-3 muscular slips (typically ribs 4-6) in the anterior axillary line. The local anaesthetic will be prepared according to body weight and a dose of 0.375% of chirocaine will be used with the addition of 1:200000 adrenaline and 1 microgram/kg of clonidine.

Group 2 - Serratus Plane Block Group

The second group will receive a serratus plane block and wound infiltration as described below:

The serratus plane block will be conducted by injecting 50% of the total available chirocaine 0.375% with adrenaline and clonidine (20mls) deep to serratus anterior under direct observation. Infiltration will be delivered into 2-3 muscular slips (typically ribs 4-6) in the anterior axillary line. The remaining 50% of local anaesthetic (20mls) will be administered by wound infiltration around the drain sites and axillary wound if present along with a 20ml 0.9% saline injection.

For clarity, please see the table summary below detailing the volumes and locations of local anaesthetic and saline injections in both groups:

20ml local anaesthetic delivered as a serratus block 20ml Saline delivered deep to serratus anterior 20ml local anaesthetic and 20ml saline wound and drain site infiltration 40ml local anaesthetic wound and drain site infiltration Control Group X √ X √ Serratus Group √ X √ X

The purpose of the saline injections is to blind the trial to the surgeon delivering the serratus block.

The anaesthesia for all patients in both groups will be induced using a combination of 0.25mg/kg ketamine, propofol and fentanyl according to standard anaesthetic protocol. All patients will receive 10mg IM morphine intraoperatively. All patients will have regular simple analgesia such as paracetamol and ibuprofen and PRN opiates (tramadol 50-100mg PRN 8 hourly) prescribed for post-operative adjunct pain management.

Patients will be blinded to which group they are randomly allocated to. Written consent and information sheets will be provided to patients and a letter sent to their GP confirming participation in the study.

Data on pain scores and the use of analgesia in recovery, the use of analgesia overnight, the presence of nausea and the pain score and mobilisation status one day after the operation will be collected. The pain score will be assessed using a standard numerical rating scale from 0-10 to score their pain subjectively where:

* 0 = No Pain
* 1-3 = Mild Pain (interferes a little with activities of daily living)
* 4-6 = Moderate Pain (interferes significantly with activities of daily living)
* 7-10 = Severe Pain (unable to perform activities of daily living)

Patients will also be followed up and one week and 3 months after their surgery to determine their recovery and the presence of any pain. This data will be collected using the FACT - B: Quality of Life Assessment 1 questionnaire.

All collected data will only be stored on NHS trust computer systems.

ELIGIBILITY:
Inclusion Criteria:

* Patients who undergo mastectomy +/- sentinel node biopsy +/- axillary clearance +/- implant reconstruction will be eligible for the study

Exclusion Criteria:

* Patients under the age of 18.

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Dates: Start 2015-10; Primary Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
To assess the serratus plane block's effectiveness in the management of post operative pain following mastectomy when compared to wound infiltration alone | 18 months

SECONDARY OUTCOMES:
To determine the proportion of patients receiving a serratus plane block during mastectomy who go on to develop chronic pain syndromes compared to patients receiving wound infiltration alone | 18 months